CLINICAL TRIAL: NCT07119736
Title: The Effects of Relaxation Using Virtual Reality in Forensic Psychiatric Patients. A Randomized Cross-over Clinical Trial
Acronym: VRelax-TAU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ONZ-2023-0315
Record Dates: First submitted 2025-07-15; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Relaxation
Keywords: stress; relaxation; virtual reality

STUDY DESIGN:
Intervention Model Description: 2 groups, 2 periods, 2 relaxation types, forensic psychiatric patients
Masking Description: participant data will be pseudonymized
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Relaxation sessions groep 1 (Experimental): there will be 10 sessions of VR and 10 sessions of standard relaxation
  Interventions: Device: VR relaxation; Other: Standard relaxation
- Relaxation sessions groep 2 (Experimental): there will be 10 sessions of standard relaxation and 10 sessions of VR
  Interventions: Device: VR relaxation; Other: Standard relaxation

INTERVENTIONS:
Device: VR relaxation — Relaxation with a VR glass and 360° video's of nature
Other: Standard relaxation — Relaxation with music, reading a book, playing computer game

SUMMARY:
During this clinical Cross-over study, the investigators want to investigate whether the use of Virtual Reality (VR) is a valuable application to achieve relaxation in forensic psychiatric patients.

This study investigates the short- and medium-term effect of VRelax on both acute and chronic stress and compares it with a standard relaxation exercise of choice (TAU).

DETAILED DESCRIPTION:
During this clinical Cross-over study, it will be investigated whether the use of Virtual Reality (VR) is a valuable application to achieve relaxation in forensic psychiatric patients within the PC Sint-Jan Baptist, Zelzate, Belgium. Due to the fact that very realistic situations can be created in VR environments that forensic psychiatric patients normally cannot experience due to their limited freedom, it seems to be an extra important asset for them that meets the limitations of confinement and freedom-restricting measures. In addition, the highly immersive character of the application supports patients who are unable to perform a standard relaxation exercise through their own imagination or empathy.

This study investigates the short- and medium-term effect of VRelax on both acute and chronic stress and compares it with a standard relaxation exercise of choice (TAU).

The relaxation software that that will be used in the study is VRelax (www.vrelax.com), which is available in Dutch (and English) for which the results of a first crossover randomized controlled trial was recently published.

The research design is a crossover randomized controlled trial with two parts: a standard relaxation of choice and a VR relaxation using the VRelax software. The VRelax app contains 360˚ VR videos of relaxing natural environments. The variety of landscapes includes beaches, mountains, proximity to animals, etc. Interactive elements are embedded in the videos, for example a game of popping air bubbles underwater, shooting stars in a night sky and audio tracks of relaxation exercises.

The study population consists of forensic psychiatric patients (depressive disorder, bipolar disorder, anxiety disorder or psychotic disorder, borderline, antisocial disorder,… (DSM-5 diagnosis)) who reside in the Sint-Jan Baptist psychiatric hospital in Zelzate, Belgium.

Before the start of the study, each candidate will be invited to an introductory session with VR to see if the person is not participating in VR disease and to make sure that the patient is still willing to participate. After consent, a baseline measurement is performed by the patient during 20 minutes, for the physical parameters using the Embrace plus device (see below).

The study will consist of 2 blocks of 10 sessions: 1 block with and 1 block without VR. Each individual is his own control in this way. Both the control measurement as the VR measurements are done in the VR room, sitting, during 20 min. The control measurement is a relaxation of choice eg. reading a book, listening to music, watching a movie, body scan, play a computer game ... The choice of relaxation form wille be registrated each session. Each block of 10 sessions must be completed within 3 the investigatorseks per patient, follothe investigatorsd by a month of rest and then the 2nd block of relaxation sessions must also be completed within 3 the investigatorseks. Each patient will therefore have 3 to 5 relaxation sessions per the investigatorsek during the study.

The VR measurement will be conducted using VRelax, which has one or more 360° videos of your choice. Only the guided meditation sessions are not used as the eyes have to be closed for that. The choice of videos per session is recorded.

Before and after each session, stress is measured via VAS scores for stress/tension and happiness on paper. At the beginning and end of each block of 10 sessions, the general stress state is measured via the "perceived stress scale" questionnaire on paper and will take 5 minutes to fill in. After the last session of each block, there is also a structured qualitative interview about the user experiences which will take 15 minutes of time.

Some physical parameters are also measured during each relaxation session via an Embrace Plus device (www.Empatica.com). These are heart rate, heart rate variability (HRV), respiratory rate, skin conductance and skin temperature.

ELIGIBILITY:
Inclusion Criteria:

* Be admitted for at least 4 months as a forensic psychiatric patient within medium or high security, at Sint-Jan Baptist in Zelzate.

Exclusion Criteria:

* Acute psychosis, acute mania, epilepsy, pacemaker, balance disorders, individuals in the acute withdrawal phase of substance or alcohol abuse, severe cardiac abnormalities, serious eye disorders, pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-10-24 (Actual); Study Completion 2024-10-24 (Actual)

PRIMARY OUTCOMES:
Difference in VAS Score for relaxation | 20 minutes
  on a scale of 1-10 How relaxed are you feeling at this moment?

SECONDARY OUTCOMES:
Difference in VAS Score for cheerfullness | 20minutes
  on a scale from 1-10 how cheerfull do you feel at this moment?

CONTACTS AND LOCATIONS:
Overall Officials: Kurt Audenaert, Prof, Principal Investigator — University Hospital, Ghent
Locations (1):
- PC Sint-Jan Baptist, Zelzate, Belgium

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-10): https://cdn.clinicaltrials.gov/large-docs/36/NCT07119736/Prot_SAP_000.pdf